CLINICAL TRIAL: NCT05659056
Title: Neoadjuvant Treatment of Pyrotinib in Combination With Trastuzumab and Abraxane in Patients With HER2-enriched Early or Locally Advanced Breast Cancer, a Single, One Arm, Multicenter II Phase Study
Brief Title: Neoadjuvant Study With Pyrotinib and Trastuzumab and Abraxane in Patients With HER2-enriched Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Shui Wang, Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NJMU-BC01
Record Dates: First submitted 2022-12-02; First posted 2022-12-21 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
Keywords: HER2-enriched, Pyrotinib, neoadjuvant therapy, pCR
MeSH Terms: conditions — Breast Neoplasms; Pathologic Complete Response | interventions — pyrotinib; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pyrotinib, trastuzumab, paclitaxel-albumin (Experimental)
  Interventions: Drug: Pyrotinib, trastuzumab, paclitaxel-albumin

INTERVENTIONS:
Drug: Pyrotinib, trastuzumab, paclitaxel-albumin — pyrotinib: 400mg orally daily; trastuzumab: 8mg/kg iv load followed by 6mg/kg iv 3-weekly for a total of 6 cycles; paclitaxel-albumin: 260mg/m2, every 3 week, a total of 6 cycles

SUMMARY:
Breast cancer is kind of highly heterogeneous tumor. The patients with the same stage and with the same treatment regimen, their prognosis varies greatly, mainly due to the different phenotypes of breast cancer and different sensitivities to drug therapy. PMA50 and BluePrint classification divides breast cancer into other inherent subtypes: Luminal A, Luminal B, HER2-enriched (HER2-E) and Basal-like. Previous studies have shown that these patients with inherent subtype of HER2-enriched are more likely to obtain higher pCR after anti-HER2 therapy. And more study and meta analysis had demonstrated the higher pCR is closely related to EFS. The genetic and molecular typing of breast cancer is closely related to the prognosis of breast cancer, so it is imperative to seek a new treatment regimen for precision treatment and maximize the therapeutic benefit of HER2-enriched patients.

ELIGIBILITY:
Inclusion Criteria:

1. female patients, 18 years ≤ age ≤ 75 years；
2. Performance Status- Eastern Cooperative Oncology Group (ECOG) 0-1
3. Histologically confirmed invasive breast cancer（early stage or locally advanced）
4. HER2 positive (HER2+++ by IHC or FISH+), and the HER2-enriched subtype screened by BulePrint test;
5. Primary breast cancer;
6. Known hormone receptor status.
7. The organs are functioning normally, like the liver function, the renal function， and the baseline left ventricular ejection fraction (LVEF)≥55% measured by ECHO
8. Signed informed consent form (ICF)

Exclusion Criteria:

1. metastatic disease (Stage IV) or inflammatory breast cancer
2. Previous or current history of malignant neoplasms, except for curatively treated:Basal and squamous cell carcinoma of the skin,Carcinoma in situ of the cervix.
3. Clinically relevant cardiovascular disease:Known history of uncontrolled or symptomatic angina, clinically significant arrhythmias, congestive heart failure, transmural myocardial infarction, uncontrolled hypertension ≥180/110);
4. A history of allergy to the drugs in this study；
5. Unable or unwilling to swallow tablets

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2022-11-29 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Pathological Complete Response (pCR) at the Time of Surgery evaluated by the investigators | Approximately 5 months from randomization following surgery or early withdrawal, whichever occurred first (Surgery was performed within 4 weeks after Cycle 6, each cycle is 21 days)
  pCR

SECONDARY OUTCOMES:
Event-free survival | Following surgery until year 2
  EFS
Objective Response Rate | Baseline up to cycle 6 (assessed at Baseline, at the time of pre-surgery), up to approximately 5 months after neoadjuvant (each cycle is 21 days)
  ORR
minimal residual lesions | Following surgery until year 2
  MRD

CONTACTS AND LOCATIONS:
Locations (1):
- JiangSu Province Hospital/ The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China